CLINICAL TRIAL: NCT00003891
Title: A Phase I Study of NX211 Given as an IV Infusion Days 1, 2 and 3 Every 3 Weeks in Patients With Solid Tumors
Brief Title: Lurtotecan Liposome in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Nexstar Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I123; CAN-NCIC-IND123 (Other: PDQ); NEXSTAR-110-02 (Other: Nexstar); CDR0000067060 (Other: PDQ)
Record Dates: First submitted 2000-06-02; First posted 2004-06-17 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: lurtotecan liposome

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of lurtotecan liposome in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) and the future dose of lurtotecan liposome in patients with advanced solid tumors. II. Assess the toxicity and pharmacokinetics of this treatment regimen in this patient population. III. Assess the response to this regimen by patients with measurable disease.

OUTLINE: This is a dose escalation, multicenter study. Patients receive lurtotecan liposome (NX211) IV over 30 minutes on days 1, 2, and 3. Courses are repeated every 3 weeks. Treatment continues for up to 6 courses in the absence of unacceptable toxicity or disease progression. The dose of NX211 is escalated in cohorts of 3-6 patients until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed at 4 weeks and every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 20-25 patients will be accrued for this study within 12-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced solid tumors that are unresponsive to existing therapy and for which no curative therapy exists Evidence of disease other than tumor marker elevation No untreated CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AST and ALT no greater than 2.5 times ULN (no greater than 5 times ULN for liver metastases) Renal: Creatinine no greater than upper limit of normal Cardiovascular: Not specified Pulmonary: Not specified Other: No prior malignancy within past 5 years except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception No active or uncontrolled infection No other serious illness or medical condition No known hypersensitivity to systemic liposomal formulation or any drug chemically related to study drug

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No greater than 3 prior chemotherapy regimens (adjuvant and metastatic) At least 3 weeks since prior adjuvant and metastatic chemotherapy (6 weeks for nitrosoureas or mitomycin and 4 weeks for carboplatin or other experimental anti cancer drugs) and recovered At least 1 year since prior high dose chemotherapy with bone marrow or stem cell support No other concurrent chemotherapy Endocrine therapy: Prior hormonal therapy allowed No concurrent hormonal therapy Radiotherapy: No prior radiotherapy to greater than 25% of bone marrow At least 4 weeks since prior radiotherapy, except for low dose myelosupressive radiotherapy, and recovered Concurrent palliative radiotherapy allowed Surgery: Not specified Other: At least 4 weeks since prior experimental drug or anticancer therapy No other concurrent investigational or anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1999-02-25 (Actual); Primary Completion 2001-06-08 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen A. Gelmon, MD, Study Chair — British Columbia Cancer Agency
Locations (2):
- Canada (2):
  - BC Cancer Agency, Vancouver, British Columbia
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goetz AD, Hammond LA, Hao D, et al.: A phase I and pharmacokinetic (PK) study of NX211 (liposomal lurtotecan) administered weekly x 4 every 6 weeks in patients with advanced solid tumors. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-388, 2002.
- [Background] Hamilton M, Wolf J, Demetri GD, et al.: Phase I pharmacokinetics of NX211 (liposomal lurtotecan) in patients with solid tumors. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-357, 2002.
- [Result] Gelmon K, Hirte H, Fisher B, Walsh W, Ptaszynski M, Hamilton M, Onetto N, Eisenhauer E. A phase 1 study of OSI-211 given as an intravenous infusion days 1, 2, and 3 every three weeks in patients with solid cancers. Invest New Drugs. 2004 Aug;22(3):263-75. doi: 10.1023/B:DRUG.0000026252.86842.e2. PMID 15122073